CLINICAL TRIAL: NCT03990207
Title: A Prospective, Multicenter, Single-Arm, Pre-Market, Pivotal Study to Evaluate Safety and Efficacy of a Novel Motorized Spiral Enteroscope for Antegrade Enteroscopy
Brief Title: The PowerSpiral Antegrade Investigational Device Exemption (IDE) Study
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Not moving forward with the study at this time. No subject were consented or enrolled
Sponsor: Olympus Corporation of the Americas (Industry)
Collaborators: Baylor Research Institute (Other); University of Massachusetts, Worcester (Other); University of Florida (Other); AdventHealth (Other); Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-OCA-01
Record Dates: First submitted 2019-06-11; First posted 2019-06-18 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Small Bowel Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- PowerSpiral Enteroscopy System (Experimental): Subjects who have a medical indication for antegrade enteroscopy
  Interventions: Device: PowerSpiral Enteroscopy System

INTERVENTIONS:
Device: PowerSpiral Enteroscopy System — Motorized spiral enteroscopy system

SUMMARY:
To evaluate safety and efficacy

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of the PowerSpiral™ Enteroscopy System, when used in subjects undergoing antegrade (per-oral) enteroscopy of the small bowel.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 22 years of age
* Medical indication for antegrade enteroscopy
* Willing and able to provide informed consent

Exclusion Criteria:

* Any medical contraindication to standard enteroscopy
* Any test that is done as part of the standard of care that would prevent the enteroscopy from being performed for safety reasons
* Unable or unwilling to provide informed consent
* Female and of child-bearing age who is currently pregnant or planning to become pregnant within the study period
* Presence of any intra-luminal or extra-luminal foreign body in the abdominal cavity
* Any prior gastric, small bowel or colonic surgery, or implantable devices in these locations (cardiac pacemakers and non-abdominal implants are acceptable)
* Known or suspected bowel obstruction, or history of bowel obstruction
* Taking anti-platelet agents or anticoagulants (other than aspirin) within last 7 days
* Known coagulation disorder
* Known or suspected esophageal stricture or Schatzki ring
* Known gastric or esophageal varices
* Suspected perforation of the gastrointestinal (GI) tract
* Previous abdominal radiation
* Inability to tolerate general anesthesia for any reason
* Inability to tolerate endotracheal intubation
* Known need for endoscopic retrograde cholangiopancreatography (ERCP) during enteroscopy
* American Society of Anesthesiologists (ASA) Classification 4 or greater

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Rate of device related serious adverse events | 7 days
  The primary safety endpoint will compare the rate of device related serious adverse events (SAE) reported in this study to the rate of device related SAEs reported in medical literature for the Spirus Medical Endo-Ease Discovery™ SB overtube
Maximum depth of endoscope insertion | Intraoperative
  The primary efficacy endpoint will compare the maximum depth of enteroscope insertion for the study device to the maximum depth of enteroscope insertion data reported in medical literature for the Spirus Medical Endo-Ease Discovery™ SB overtube.

SECONDARY OUTCOMES:
Total procedure time | Intraoperative
  Measured from initial enteroscope introduction through the bite block to final enteroscope withdrawal through the bite block in minutes.
Insertion time | Intraoperative
  Measured from the initial enteroscope introduction through the bite block to maximum depth of enteroscope insertion measured in minutes
Withdrawn time | Intraoperative
  Measured from maximum depth of enteroscope insertion excluding any time spent on therapeutic interventions, to final enteroscope withdrawal through bite block measured in minutes.
Total enteroscopy rate | Intraoperative
  Percentage of subjects where the entire small intestine is intubated with the enteroscopy from pylorus to cecum.
Diagnostic yield | Intraoperative
  Percentage of subjects where enteroscopy produces the findings required to establish diagnosis.
Adverse events | 7 days post-procedure
  SAEs regardless of relationship to study device and/or procedure, and non-SAEs related to study device and/or procedure
Device deficiencies | Intraoperative
  Number of device deficiencies during the enteroscopy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Daniel DeMarco, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Olympus Corporation of the Americas, Southborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baniya R, Upadhaya S, Subedi SC, Khan J, Sharma P, Mohammed TS, Bachuwa G, Jamil LH. Balloon enteroscopy versus spiral enteroscopy for small-bowel disorders: a systematic review and meta-analysis. Gastrointest Endosc. 2017 Dec;86(6):997-1005. doi: 10.1016/j.gie.2017.06.015. Epub 2017 Jun 23. PMID 28652176
- [Background] Buscaglia JM, Richards R, Wilkinson MN, Judah JR, Lam Y, Nagula S, Draganov PV. Diagnostic yield of spiral enteroscopy when performed for the evaluation of abnormal capsule endoscopy findings. J Clin Gastroenterol. 2011 Apr;45(4):342-6. doi: 10.1097/MCG.0b013e3181eeb74b. PMID 20861800
- [Background] Khashab MA, Lennon AM, Dunbar KB, Singh VK, Chandrasekhara V, Giday S, Canto MI, Buscaglia JM, Kapoor S, Shin EJ, Kalloo AN, Okolo PI 3rd. A comparative evaluation of single-balloon enteroscopy and spiral enteroscopy for patients with mid-gut disorders. Gastrointest Endosc. 2010 Oct;72(4):766-72. doi: 10.1016/j.gie.2010.04.043. Epub 2010 Jul 8. PMID 20619404
- [Background] Akerman PA, Haniff M. Spiral enteroscopy: prime time or for the happy few? Best Pract Res Clin Gastroenterol. 2012 Jun;26(3):293-301. doi: 10.1016/j.bpg.2012.03.008. PMID 22704571